CLINICAL TRIAL: NCT07309341
Title: Effects of Isotretinoin on Nasal Mucociliary Clearance and Olfactory Function
Brief Title: Effects of Isotretinoin on Smell
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ISO51116; 1919B012412359 (Other Grant/Funding Number: This study was supported by the Scientific and Technological Research Council of Turkey (TÜBİTAK).)
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Smell Dysfunction
Keywords: olfaction; smell disfunction; isotretinoin
MeSH Terms: conditions — Olfaction Disorders; Anosmia | interventions — Isotretinoin

STUDY DESIGN:
Masking Description: The statistician responsible for analyzing the olfactory test scores and questionnaire data will be masked to the timepoint (baseline vs post-treatment) and participant information. Clinical investigators and participants are not masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isotretinoin Treatment Group (Experimental): Participants in this arm will receive standard-of-care oral isotretinoin prescribed by the Dermatology Department for the treatment of acne vulgaris. The dosage and duration of isotretinoin therapy will follow routine clinical practice and will be determined by the treating dermatologist. Olfactory function and nasal symptom assessments will be performed before starting isotretinoin and after at least four weeks of treatment.
  Interventions: Drug: isotretinoin

INTERVENTIONS:
Drug: isotretinoin — Oral isotretinoin prescribed as standard-of-care treatment for acne vulgaris. The dosage, formulation, and duration of therapy will follow routine clinical practice and will be determined by the treating dermatologist based on the participant's clinical condition and body weight. Participants will typically receive daily oral isotretinoin for at least four weeks before the post-treatment assessments.

SUMMARY:
Isotretinoin is a common medicine used to treat moderate to severe acne. It often causes dryness of the skin and the inside of the nose. Because a normal sense of smell depends on a healthy nasal lining, this dryness may affect how well a person can smell.

This study will examine whether isotretinoin treatment changes the sense of smell in adults with acne. Before starting isotretinoin, participants will complete a standardized smell test and two short questionnaires about nasal symptoms and quality of life (NOSE and SNOT-22). After at least 4 weeks of treatment, the same smell test and questionnaires will be repeated.

By comparing results before and after treatment, the study will test the hypothesis that isotretinoin has a negative effect on olfactory function and may reduce patients' ability to smell.

DETAILED DESCRIPTION:
Isotretinoin is a systemic retinoid widely used for the treatment of moderate to severe acne that does not respond adequately to conventional topical or oral therapies. Although highly effective, isotretinoin is known to cause mucocutaneous dryness, which may alter the nasal environment and potentially influence olfactory function. The sense of smell depends on the integrity of the olfactory epithelium, the moisture of the nasal mucosa, and the ability of odorant molecules to reach and dissolve within the mucus layer. Changes in these factors may lead to measurable reductions in olfactory sensitivity or identification ability.

Previous studies examining the effects of isotretinoin on olfaction have produced conflicting results. One investigation reported an increase in olfactory sensitivity during treatment, while another found a decrease in smell function using a different testing method. These inconsistent findings, combined with the limited number of available studies, highlight the need for further research using standardized and reproducible assessment tools.

This prospective clinical study will evaluate olfactory function in adults initiating isotretinoin therapy for dermatologic indications. Participants will undergo a structured olfactory assessment using the Connecticut Chemosensory Clinical Research Center (CCCRC) smell test, which includes both odor identification and discrimination components. In parallel, patient-reported nasal symptoms and sinonasal-related quality of life will be assessed using the NOSE and SNOT-22 questionnaires, allowing a broader understanding of subjective nasal changes that may accompany isotretinoin use.

All assessments will be performed at two time points: before the start of isotretinoin therapy and after a minimum of four weeks of continuous treatment. This within-subject design will allow comparison of pre-treatment and post-treatment measurements to determine whether isotretinoin produces quantifiable changes in olfactory performance. The study hypothesis is that isotretinoin may negatively affect olfactory function due to its well-recognized drying effects on the nasal mucosa.

The findings of this research may assist clinicians in counseling patients regarding potential sensory side effects of isotretinoin and may provide a basis for further investigations into the mechanisms by which systemic medications influence nasal physiology and smell perception.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acne and scheduled to start oral isotretinoin as part of routine dermatology care
* Willing to participate and able to give informed consent
* Not currently smoking
* No history of allergic rhinitis, sinusitis, or active upper respiratory infection
* No medical condition known to affect the sense of smell

Exclusion Criteria:

* Younger than 18 years or older than 45 years
* Current cigarette smoking
* History of chronic sinonasal disease
* Any condition that would prevent completing the smell test
* Not willing to continue participation or withdrawal of consent at any time

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Olfactory Function Score | Baseline and 4 weeks after starting isotretinoin treatment.
  Change in olfactory function from baseline to at least 4 weeks after initiation of oral isotretinoin therapy, measured using the Connecticut Chemosensory Clinical Research Center (CCCRC) smell test. The CCCRC test includes odor identification and odor discrimination components, and yields a composite score representing overall olfactory performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Uşak University Faculty of Medicine, Uşak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because institutional policy does not permit external sharing of health-related data.